CLINICAL TRIAL: NCT05036304
Title: Supporting Aging Through Green Exercise (SAGE): Comparing the Cognitive Effects of Outdoor Versus Indoor Exercise Among Older Adults With Mild Cognitive Impairment
Brief Title: Supporting Aging Through Green Exercise (SAGE)
Acronym: SAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Teresa Liu-Ambrose, Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H21-00406
Record Dates: First submitted 2021-09-01; First posted 2021-09-05 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Mild Cognitive Impairment; Aging
Keywords: green space; cognitive function; aerobic exercise
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Assessor will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Exercise Indoors (Active Comparator): Each session will consist of 10 min of warm-up, 40 min of aerobic exercise, and 10 min of cool-down. Aerobic exercise will be progressive and of moderate intensity. During training, each participant will wear a heart rate monitor and will be asked to work initially at approximately 45% of his/her target heart rate (i.e., heart rate reserve (HRR)) and gradually progress to reach the target of 70% of HRR over the 12-week study period. Participants will also subjectively monitor workout intensity using the 20-point Borg's Rating of Perceived Exertion. Participants will walk or jog on treadmills or cycle on stationary bikes in the Exercise Prescription Suite of the Centre for Hip Health and Mobility.
  Interventions: Other: Aerobic Exercise Indoors
- Aerobic Exercise Outdoors (Experimental): Each session will consist of 10 min of warm-up, 40 min of aerobic exercise, and 10 min of cool-down. Aerobic exercise will be progressive and of moderate intensity. During training, each participant will wear a heart rate monitor and will be asked to work initially at approximately 45% of his/her target heart rate (i.e., heart rate reserve (HRR)) and gradually progress to reach the target of 70% of HRR over the 12-week study period. Participants will also subjectively monitor workout intensity using the 20-point Borg's Rating of Perceived Exertion. participants will walk or jog pre-determined routes in trails of an urban forest (Pacific Spirit Park).
  Interventions: Other: Aerobic Exercise Outdoors

INTERVENTIONS:
Other: Aerobic Exercise Indoors — Each session will consist of 10 min of warm-up, 40 min of aerobic exercise, and 10 min of cool-down. Aerobic exercise will be progressive and of moderate intensity. During training, each participant will wear a heart rate monitor and will be asked to work initially at approximately 45% of his/her target heart rate (i.e., heart rate reserve (HRR)) and gradually progress to reach the target of 70% of HRR over the 12-week study period. Participants will also subjectively monitor workout intensity using the 20-point Borg's Rating of Perceived Exertion. Participants will walk or jog on treadmills or cycle on stationary bikes in the Exercise Prescription Suite of the Centre for Hip Health and Mobility.
  Arms: Aerobic Exercise Indoors
Other: Aerobic Exercise Outdoors — Each session will consist of 10 min of warm-up, 40 min of aerobic exercise, and 10 min of cool-down. Aerobic exercise will be progressive and of moderate intensity. During training, each participant will wear a heart rate monitor and will be asked to work initially at approximately 45% of his/her target heart rate (i.e., heart rate reserve (HRR)) and gradually progress to reach the target of 70% of HRR over the 12-week study period. Participants will also subjectively monitor workout intensity using the 20-point Borg's Rating of Perceived Exertion. Participants will walk or jog pre-determined routes in trails of an urban forest (Pacific Spirit Park)
  Arms: Aerobic Exercise Outdoors

SUMMARY:
Aerobic exercise is an evidence-based approach to mitigate cognitive decline in older adults with mild cognitive impairment (MCI). Emerging evidence suggests that the cognitive benefits of exercise may be enhanced when performed in outdoor, natural settings, as compared to indoor or built settings. Thus, the investigators aim to compare the effects of outdoor versus indoor walking programs on cognitive function among older adults with MCI. Secondary outcomes are motor function, emotional well-being, health-related behaviours, and quality of life. Participants will be randomly assigned to a 12--week, 3x/week program of either outdoor walking on forest trails or indoor walking on a treadmill. A 3-month followup will also be completed after trial completion.

DETAILED DESCRIPTION:
Study Design: A 12-week, single-blinded, trial with two experimental arms. Participants will be randomized (1:1) to either outdoor walking (OP) or indoor walking or cycling (IP). Measurement will occur in person at baseline and at trial completion. Additionally, follow-up measurement of questionnaire-based outcomes will occur via email or phone at 3 months following trial completion. Outcome assessors will be trained by the research team and blinded to group allocation of the participants.

Participants: 68 community-dwelling adults aged 65-80 years old with probable MCI and in sufficient health to participate in aerobic exercise of moderate intensity

Interventional Arms: All participants will receive three group-based training sessions per week for 12 weeks, under the supervision of instructors with a relevant background and first aid certification. Each session will consist of 10 min of warm-up, 40 min of aerobic exercise, and 10 min of cool-down. For both OP and IP, aerobic exercise will be progressive and of moderate intensity. During training, each participant will wear a heart rate monitor and will be asked to work initially at approximately 45% of their heart rate reserve (HRR) and gradually progress to reach the target of 70% of HRR over the 12-week study period. Participants will also subjectively monitor workout intensity using the 20-point Borg's Rating of Perceived Exertion. OP participants will walk or jog a pre-determined route in trails of an urban forest (Pacific Spirit Park). IP participants will walk or jog on treadmills in the Exercise Prescription Suite of the Centre for Hip Health and Mobility (CHHM). Both OP and IP training groups will have a participant to instructor ratio of 3:1. To promote adherence to the exercise program, sessions will be offered at times that are convenient for each individual participant. Protocols will be adjusted as necessary to align with COVID-19 guidelines.

Measurement of descriptors and outcomes: Standardized protocols will be developed and study personnel will be trained. Assessors will be blinded to treatment allocation. We will measure descriptors and outcomes at baseline and at trial completion. Each measurement session will be 2 hours in duration. For these measurements, participants will complete a session of behavioural and clinical testing at the VCH Research Pavilion and the CHHM. To account for time-of-day effects, each participant's session start time will be the same at both timepoints, and the order of the assessments will be the same for all participants.

ELIGIBILITY:
Inclusion Criteria:

1. achieve a score ≥18/30 and ≤24/30 on the Montreal Cognitive Assessment
2. have subjective cognitive impairment based on interview
3. have no significant impairment in daily function, as determined by a score ≥6/8 on the Lawton and Brody Instrumental Activities of Daily Living Scale
4. no diagnosis of dementia
5. aged 65 to 80 years old
6. live independently in their own home
7. live in the Greater Vancouver area
8. read, write, and speak English with acceptable visual and auditory acuity
9. are cleared to start a supervised exercise programme based on the Physical Activity Readiness Questionnaire for Everyone
10. able to walk independently
11. able to provide informed consent

Exclusion Criteria:

1. participating in regular moderate to vigorous intensity aerobic exercise in the last 3 months
2. planning to enroll in a concurrent exercise or drug trial targeting cognitive function
3. diagnosed with a neurological, cerebrovascular, or psychiatric disease, or other chronic medical condition requiring intensive treatment and monitoring
4. have major impairments in eyesight, hearing or motor movements
5. have clinically significant neuropathy or musculoskeletal or joint disease
6. have a recent traumatic brain injury, including concussions
7. are currently using prescribed cognitive intervention or electromagnetic stimulation
8. at the time of recruit, indicate they recently (within the last 2 months) or will start taking drugs that significantly alter cognition, movement, or affect, such as cholinesterase inhibitors, anticholinergics, hormone replacement therapy, or antidepressants

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
Change in List Sorting Performance | Baseline to 12 weeks
  This is a measure of working memory
Change in Digits Span Forwards and Backwards | Baseline to 12 weeks
  This is a measure of working memory.

SECONDARY OUTCOMES:
Change in NIH Toolbox Cognitive Battery Performance | Baseline to 12 weeks
  Measures different cognitive domains, with a focus on executive functions
Change in Digit Symbol Substitute Test | Baseline to 12 weeks
  A measure of processing speed and executive functions.
Change in the Short Physical Performance Battery | Baseline to 12 weeks
  A measure of balance and mobility
Change in Timed Up and Go Test | Baseline to 12 weeks
  A measure of general mobility
Change in State-Trait Anxiety Inventory | Baseline to 12 weeks and 6 months
  A measure of anxiety
Change in Centre for Epidemiological Studies Depression Scale | Baseline to 12 weeks and 6 months
  A measure of depressive symptoms
Change in Blood Pressure | Baseline to 12 weeks
  Systolic and diastolic blood pressure
Change in sensor measured sleep | Baseline to 12 weeks
  Using MotionWatch 8 to measure sleep quality
Change in sensor measured physical activity | Baseline to 12 weeks
  Using MotionWatch 8 to measure levels and amount of physical activity
Change in Physical Activity Scale for the Elderly | Baseline to 12 weeks and 6 months
  A self-report measure of physical activity, higher scores indicate higher activity
Change in Pittsburgh Sleep Quality Index | Baseline to 12 weeks and 6 months
  A self-report measure of sleep quality, higher scores indicate poorer sleep quality
Change in ICEpop CAPability measure for Older people (ICECAP-O) | Baseline to 12 weeks and 6 months
  A measure of quality of life, higher values indicate better quality of life
5-level EuroQoL 5-dimension (EQ-5D-5L) questionnaire | Baseline to 12 weeks and 6 months
  A measure of quality of life, higher values indicate better quality of life
Change in gait speed, derived from Short Physical Performance Battery | Baseline to 12 weeks.
  A measure of walking speed.
Changes in hemodynamics of the brain as measured by fNIRS during the N-Back Task | Baseline to 12 weeks.
  A measure of brain function.
Changes in Feeling Scale | Baseline to 12 weeks.
  Measure of affective valence
Changes in Exercise Enjoyment Scale | Baseline to 12 weeks.
  An affective measure
Changes in Felt Arousal Scale | Baseline to 12 weeks
  Measure of affective activation

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Liu-Ambrose, PhD, Principal Investigator — University of British Columbia; Matthew Noseworthy, BSc, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada